CLINICAL TRIAL: NCT00983606
Title: An Observational Prospective Study to Assess Respiratory Syncytial Virus (RSV) Respiratory Events Among Premature Infants (32 to 35 Week Gestational Age) - Outcomes and Risk Tracking Study (The Report Study)
Brief Title: An Observational Study to Assess Respiratory Syncytial Virus (RSV) Respiratory Events Among Premature Infants
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MI-MA213
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum (frozen)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: 32 to 35 WGA Infants less than six months of age by RSV season peak.

SUMMARY:
The primary objective is to assess the burden of respiratory disease in outpatient settings among 32 to 35 weeks' gestational age (wGA) infants in the USA who did not receive RSV prophylaxis during the infants' first RSV season.

DETAILED DESCRIPTION:
The primary objective is to determine the burden of RSV disease in outpatient settings among 32 to 35 wGA infants in the USA who did not receive RSV prophylaxis, as measured by rate of RSV-associated outpatient lower respiratory tract illness (LRI) during the infants' first RSV season.

ELIGIBILITY:
Inclusion Criteria:

* Premature at birth (from 32 weeks and 0 days to 35 weeks and 6 days GA)
* Age 6 months or less at the time of screening, and born in May 2009 through January 2010 for Season 1, or May 2010 through February 2011 for Season 2
* Written informed consent and any locally required authorization (eg, HIPAA), obtained from the subject's parent/or guardian prior to performing any protocol-related procedures.

Exclusion Criteria:

* Receipt of any RSV prophylactic agent: at any time prior to study participation
* Participation in studies of investigational RSV prophylaxis or RSV therapeutic agents
* Presence of bronchopulmonary dysplasia,hemodynamically significant congenital heart disease, congenital neuromuscular or congenital airway defects
* Any condition that, in the opinion of the investigator, would limit life expectancy to less than 6 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Premature babies at birth - (32-35 WGA)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence rate of outpatient RSV LRI during the RSV season, with RSV LRI determined by real time RT-PCR | Sep. 2009-Feb. 2010; Sep. 2010-Feb. 2011

SECONDARY OUTCOMES:
Rate of RSV-associated emergency department (ED) visits during the RSV season | 2009-2010; 2010- 2011
Rate of RSV-associated hospitalization during the RSV season | 2009-2010; 2010-2011
Rate of risk factors for RSV-associated outpatient LRI, hospitalization, and ED visits | 2009-2010; 2010-2011
Rate of risk factors for RSV infection | 2009-2010; 2010-2011

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Groothuis, MD, Study Director — MedImmune LLC
Locations (199):
- United States (199):
  - Research Site, Birmingham, Alabama
  - Research Site, Dothan, Alabama
  - Research Site, Greenville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Prattville, Alabama
  - Research Site, Scottsboro, Alabama
  - Research Site, Selma, Alabama
  - Research Site, Sylacauga, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Prescott, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Benton, Arkansas
  - Research Site, Bentonville, Arkansas
  - Research Site, Fort Smith, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site, Chico, California
  - Research Site, Fountain Valley, California
  - Research Site, Fresno, California
  - Research Site, Granada Hills, California
  - Research Site, Hollister, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, National City, California
  - Research Site, San Diego, California
  - Research Site, San Jose, California
  - Research Site, Santa Ana, California
  - Research Site, Ventura, California
  - Research Site, Aurora, Colorado
  - Research Site, Centennial, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, Longmont, Colorado
  - Research Site, Louisville, Colorado
  - Research Site, Newark, Delaware
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Cantonment, Florida
  - Research Site, Cocoa Beach, Florida
  - Research Site, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lake Mary, Florida
  - Research Site, Merritt Island, Florida
  - Research Site, Miami, Florida
  - Research Site, New Port Richey, Florida
  - Research Site, Orange Park, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Alpharetta, Georgia
  - Research Site, Clarkston, Georgia
  - Research Site, College Park, Georgia
  - Research Site, Hinesville, Georgia
  - Research Site, Jesup, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Royston, Georgia
  - Research Site, Snellville, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Crystal Lake, Illinois
  - Research Site, Evergreen Park, Illinois
  - Research Site, Libertyville, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site, New Albany, Indiana
  - Research Site, Sellersburg, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Dubuque, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Bardstown, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Somerset, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Brockton, Massachusetts
  - Research Site, Framingham, Massachusetts
  - Research Site, Pittsfield, Massachusetts
  - Research Site, Westford, Massachusetts
  - Research Site, Woburn, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bingham Farms, Michigan
  - Research Site, Niles, Michigan
  - Research Site, Stevensville, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Brookhaven, Mississippi
  - Research Site, Jackson, Mississippi
  - Research Site, Newton, Mississippi
  - Research Site, Bridgeton, Missouri
  - Research Site, Joplin, Missouri
  - Research Site, North Kansas City, Missouri
  - Research Site, Saint Joseph, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Butler, New Jersey
  - Research Site, Neptune City, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, Princeton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Vineland, New Jersey
  - Research Site, Woodcliff Lake, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Commack, New York
  - Research Site, Jamaica, New York
  - Research Site, Jericho, New York
  - Research Site, Liverpool, New York
  - Research Site, Mineola, New York
  - Research Site, Nanuet, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Utica, New York
  - Research Site, Valley Stream, New York
  - Research Site, Albemarle, North Carolina
  - Research Site, Asheville, North Carolina
  - Research Site, Boone, North Carolina
  - Research Site, Clyde, North Carolina
  - Research Site, Morganton, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Raliegh, North Carolina
  - Research Site, Trinity, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Coal Grove, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Fairfield, Ohio
  - Research Site, Huber Heights, Ohio
  - Research Site, Kent, Ohio
  - Research Site, Lancaster, Ohio
  - Research Site, Massillon, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Youngstown, Ohio
  - Research Site, Norman, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Grants Pass, Oregon
  - Research Site, Gresham, Oregon
  - Research Site, McMinnville, Oregon
  - Research Site, Hanover, Pennsylvania
  - Research Site, Kittanning, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Barnwell, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Cheraw, South Carolina
  - Research Site, Clarksville, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Lebanon, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Carrollton, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Smithville, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tomball, Texas
  - Research Site, St. George, Utah
  - Research Site, West Jordan, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Chesapeake, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Glen Allen, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Springfield, Virginia
  - Research Site, Vienna, Virginia
  - Research Site, Centralia, Washington
  - Research Site, Spokane, Washington
  - Research Site, Woodinville, Washington
  - Research Site, Charleston, West Virginia
  - Research Site, La Crosse, Wisconsin
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Monroe, Wisconsin

REFERENCES:
- [Derived] Simoes EA, Anderson EJ, Wu X, Ambrose CS. Effects of Chronologic Age and Young Child Exposure on Respiratory Syncytial Virus Disease among US Preterm Infants Born at 32 to 35 Weeks Gestation. PLoS One. 2016 Nov 29;11(11):e0166226. doi: 10.1371/journal.pone.0166226. eCollection 2016. PMID 27898687
- [Derived] Ambrose CS, Anderson EJ, Simoes EA, Wu X, Elhefni H, Park CL, Sifakis F, Groothuis JR. Respiratory syncytial virus disease in preterm infants in the U.S. born at 32-35 weeks gestation not receiving immunoprophylaxis. Pediatr Infect Dis J. 2014 Jun;33(6):576-82. doi: 10.1097/INF.0000000000000219. PMID 24622396